CLINICAL TRIAL: NCT00335829
Title: Phase II Trial of Bevacizumab Combined With Transarterial Chemoembolization (TACE) for Hepatocellular Carcinoma
Brief Title: Bevacizumab and Chemoembolization in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0598 CDR0000483104; JHOC-J0598; JHOC-NA_00001249
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; adult primary hepatocellular carcinoma; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab; Drug Therapy; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm, received bevacizumab and TACE (Experimental)
  Interventions: Biological: bevacizumab; Drug: chemotherapy; Drug: embolization therapy; Procedure: hepatic artery infusion

INTERVENTIONS:
Biological: bevacizumab
Drug: chemotherapy
Drug: embolization therapy
Procedure: hepatic artery infusion

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoembolization kills tumor cells by carrying chemotherapy drugs directly into the tumor and blocking the blood flow to the tumor. Giving bevacizumab together with chemoembolization may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with chemoembolization works in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Improve median progression-free survival of patients with unresectable hepatocellular cancer treated with bevacizumab and transarterial chemoembolization therapy.

Secondary

* Characterize the safety and toxicity of this regimen in these patients.
* Determine the response rate in patients treated with this regimen.

OUTLINE: Patients receive bevacizumab once in weeks 1, 3, and 5. Beginning in week 3, patients also receive transarterial chemoembolization (TACE) therapy. Treatment repeats approximately every 8 weeks for up to 3 courses. Patients achieving < 100% necrosis by MRI after the first course receive 2 additional courses of bevacizumab and TACE.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* hepatocellular carcinoma

  * Unresectable disease
  * Child's class A or B with liver-predominant and asymptomatic extrahepatic disease NOTE: *A highly suspicious liver mass on CT scan or MRI in the presence of alpha fetoprotein > 200 mg/dL may be used as alternative diagnostic criterion

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 50,000/mm³
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5.0 times upper limit of normal (ULN)
* Bilirubin ≤ 5.0 mg/dL
* Creatinine normal OR creatinine clearance > 50 mL/min
* No significant traumatic injury within the past 28 days
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, nonhealing wound, ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

* No major surgery or open biopsy within the past 28 days
* No minor surgery (e.g., fine-needle aspirations or core biopsies) within the past 7 days
* No chemotherapy within the past 4 weeks
* No radiotherapy within the past 21 days
* No concurrent major surgery
* No other concurrent chemotherapy
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F. Geschwind, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a diagnosis of unresectable hepatocellular carcinoma (HCC) were enrolled on this protocol to receive a combination of intravenous bevacizumab and transarterial chemoembolization (TACE) therapy. A total of 26 patients were enrolled on protocol; 10 patients at Northwestern University and 16 at Johns Hopkins University.
Groups:
- Single Arm, Received Bevacizumab and TACE: Patients received intravenous bevacizumab (10mg/kg) and chemoembolization for up to 3 cycles over 6 months. After completion of last treatment cycle, follow-up including clinic visits and imaging was performed every 8 to 12 weeks.
Period: Overall Study
Arm/Group | Single Arm, Received Bevacizumab and TACE
Started | 26
Received Bevacizumab (Patients reaching this milestone were evaluated for safety and toxicity outcomes) | 26
Received First TACE | 25 (1 patient left after receiving bevacizumab but prior to first TACE)
Completed (Patients who were evaluable for tumor response for imaging outcomes) | 23
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm, Received Bevacizumab and TACE: bevacizumab
  chemotherapy
  embolization therapy
  hepatic artery infusion
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 64 [31 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Description: This outcome was not assessed. Instead, the primary outcome of time to tumor progression (TTP) of the targeted lesions and secondary outcomes of TTP of nontargeted lesions and overall TTP were assessed and reported.
Time Frame: Time through study completion, an average of 1 year
Population: PFS analysis was not conducted. No data were collected for this Outcome Measure
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Tumor Progression (TTP) of Targeted Lesions
Description: Time to tumor progression was estimated via Kaplan-Meier methodology using the 23 patients who underwent treatment.
Time Frame: 6 months and 1 year
Measure: Number; unit: months
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
months | NA — Among the targeted lesions, the majority had no evidence of progression at 6 months (86%) or at 1 year (53%). The median TTP of the targeted lesions from the start of therapy was not reached at last follow-up of 1 year.

3. Secondary Outcome: TTP of Nontargeted Lesions Within the Liver
Description: TTP of nontargeted lesions assessed via Kaplan-Meier methodology.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
months | 9.1 [6.5 to 9.1]

4. Secondary Outcome: Overall TTP
Description: Overall TTP assessed via Kaplan-Meier methodology.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
months | 7.2 [5.8 to 9.1]

5. Secondary Outcome: TTP Rate at 6 Months and 1 Year
Description: Overall TTP assessed via Kaplan-Meier methodology at 6 months and 1 year
Time Frame: 6 months and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
percentage of participants
  TTP rate at 6 months | 65 [47 to 90]
  TTP rate at 1 year | 23 [9 to 60]

6. Secondary Outcome: Overall Survival (OS)
Description: OS assessed via Kaplan-Meier methodology both from initiation of therapy and from the date of diagnosis until death.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
months
  OS from start of therapy | 10.8 [4.8 to 24.7]
  OS from date of diagnosis | 23.6 [12.8 to 31.5]

7. Secondary Outcome: Response Rate - Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Efficacy as assessed by radiographic tumor response using RECIST criteria at baseline, 3 weeks after TACE, and 4 weeks after completion of final cycle.
  Complete Response (CR): Disappearance of all lesions targeted by therapy Partial Response (PR): At least 30% decrease in the sum of longest diameter (LD) of lesions targeted by therapy Progressive Disease (PD): At least 20% increase in sum of LD of lesions targeted by therapy Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 8
  Stable Disease (SD) | 15
  Progressive Disease (PD) | 0
  Overall response rate (CR + PR) | 8
  Disease control rate (CR + PR + SD) | 23

8. Secondary Outcome: Response Rate - Based on Tumor Enhancement
Description: Efficacy as assessed by radiographic tumor response utilizing the following tumor enhancement criteria:
  Complete Response (CR): 100% tumor necrosis of the target lesion(s) upon completion of any of the 3 cycles of TACE therapy Partial Response (PR): Greater than 50% tumor necrosis of target lesion(s) Progressive Disease (PD): Reappearance or increased tumor enhancement greater than 25% in target lesion(s) Stable Disease (SD): Cases that do not meet CR or PR and did not demonstrate evidence of tumor progression.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 23
Participants
  Complete Response (CR) | 4
  Partial Response (PR) | 10
  Stable Disease (SD) | 9
  Progressive Disease (PD) | 0
  Overall response rate (CR + PR) | 14
  Disease control rate (CR + PR + SD) | 23

9. Secondary Outcome: Safety and Treatment Toxicity - Cycle 1 Pre-TACE
Description: Safety and toxicity assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3.0) for all patients (n=26) who received bevacizumab prior to TACE therapy.
Time Frame: Cycle 1 pre-TACE - 2 weeks
Measure: Number; unit: adverse events
Units Other Than Participants: Adverse events
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 26
Number analyzed (Adverse events) | 24
adverse events
  Coagulation | 3
  Fatigue | 2
  Weight loss | 1
  Ascites | 1
  Anorexia | 1
  Nausea | 2
  Vomiting | 1
  Esophageal varices | 1
  Elevated ALT | 1
  Elevated AST | 2
  Hyperbilirubinemia | 3
  Hyponatremia | 2
  Encephalopathy | 1
  Right upper quadrant pain | 1
  Proteinuria | 1
  Respiratory | 1

10. Secondary Outcome: Safety and Treatment Toxicity - Cycle 1 Post-TACE
Description: Safety and toxicity assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3.0) for 25 who completed the first cycle of TACE and bevacizumab therapy
Time Frame: Cycle 1 post-TACE - 5 weeks
Population: 1 out of the initial 26 patients did not complete the first TACE on protocol and was not included in this assessment.
Measure: Number; unit: adverse events
Units Other Than Participants: Adverse events
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 25
Number analyzed (Adverse events) | 151
adverse events
  Anemia | 10
  Leukocytopenia | 7
  Lymphopenia | 8
  Edema | 3
  Ischemia | 1
  Coagulation | 10
  Fatigue | 12
  Night sweats | 2
  Weight loss | 6
  Ascites | 1
  Anorexia | 11
  Nausea | 4
  Vomiting | 6
  HEENT | 2
  Elevated ALT | 7
  Elevated AST | 7
  Hyperbilirubinemia | 6
  Liver failure | 1
  Cellulitis | 1
  Colangitis | 1
  Hyperglycemia | 8
  Hypocalcemia | 3
  Hypokalemia | 2
  Hyponatremia | 7
  Delirium | 1
  Psychosis | 1
  Abdominal pain, not otherwise specified (NOS) | 6
  Epigastric pain | 1
  Right upper quadrant pain | 3
  Chest pain | 2
  Pain - other | 3
  Dyspnea | 2
  Acute renal failure | 1
  Proteinuria | 2
  Respiratory | 3

11. Secondary Outcome: Safety and Treatment Toxicity - Cycles 2 and 3
Description: Safety and toxicity assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3.0) for patients (n=14) who completed 2 or 3 cycles of TACE and bevacizumab therapy
Time Frame: 6 months
Population: 14 out of the original 26 study participants completed 2 or 3 cycles of TACE and bevacizumab therapy - adverse events associated with these patients for cycles 2 and 3 assessed.
Measure: Number; unit: adverse events
Units Other Than Participants: Adverse events
Arm/Group | Single Arm, Received Bevacizumab and TACE
Number analyzed (Participants) | 14
Number analyzed (Adverse events) | 103
adverse events
  Leukocytopenia | 7
  Lymphopenia | 12
  Heart failure | 1
  Edema | 2
  Coagulation | 5
  Fatigue | 11
  Weight loss | 2
  Dermatologic | 3
  Endocrine | 2
  Ascites | 3
  Anorexia | 2
  Duodenal perforation | 1
  Nausea | 1
  Vomiting | 2
  Elevated ALT | 2
  Elevated AST | 6
  Hyperbilirubinemia | 4
  Clostridium difficile | 1
  Hyperglycemia | 11
  Hypocalcemia | 2
  Hypokalemia | 1
  Hyponatremia | 4
  Fracture | 1
  Cord compression | 1
  Stroke | 1
  Right upper quadrant pain | 4
  Pain - other | 3
  Dyspnea | 1
  Proteinuria | 2
  Respiratory | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Arm, Received Bevacizumab and TACE
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Received Bevacizumab and TACE (N=26)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Cerebral infarct (Nervous system disorders) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Esophageal varices (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Received Bevacizumab and TACE (N=26)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Leukocytopenia (Investigations) | 7 (14)
Lymphopenia (Investigations) | 12 (20)
Edema (General disorders) | 3 (5)
Coagulation/Elevated INR (Investigations) | 10 (15)
Fatigue (General disorders) | 12 (25)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Weight loss (General disorders) | 6 (8)
Dermatologic (Skin and subcutaneous tissue disorders) | 3 (3)
Endocrine (Endocrine disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 11 (14)
Nausea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 6 (9)
Elevated ALT (Investigations) | 7 (10)
Elevated AST (Investigations) | 7 (15)
Hyperbilirubinemia (Investigations) | 6 (13)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 7 (11)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Right upper quadrant pain (Gastrointestinal disorders) | 4 (8)
Chest pain (General disorders) | 2 (2)
Pain - other (General disorders) | 3 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No